CLINICAL TRIAL: NCT02112552
Title: A Pilot Phase II Trial of Intravenous Paclitaxel and Intraperitoneal Carboplatin Followed by Radiation in Patients With Advanced Stage Uterine Serous Carcinoma
Brief Title: Paclitaxel and Intraperitoneal Carboplatin Followed by Radiation Therapy in Treating Patients With Stage IIIC-IV Uterine Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual. Study formally terminated by PI on 12/1/2017
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-02-058; NCI-2013-01226 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-02-058 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Serous Adenocarcinoma; Stage IIIA Uterine Corpus Cancer; Stage IIIB Uterine Corpus Cancer; Stage IIIC1 Uterine Corpus Cancer; Stage IIIC2 Uterine Corpus Cancer; Stage IVA Uterine Corpus Cancer; Stage IVB Uterine Corpus Cancer
MeSH Terms: interventions — Paclitaxel; Taxes; Carboplatin; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel, carboplatin, radiotherapy) (Experimental): CHEMOTHERAPY: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IP on day 1. Treatment repeats every 21 days for up to 6 courses (weeks 1-18) in the absence of disease progression or unacceptable toxicity.
  RADIATION: At provider discretion, patients may undergo 3D conformal or IMRT 5 days a week for 5 weeks (weeks 19-23).
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; TAX
Drug: Carboplatin — Given IP
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D conformal radiation therapy
  Other Names: 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot, phase II trial studies the side effects and how well paclitaxel given into the vein and carboplatin given directly into the abdominal cavity (intraperitoneally) followed by radiation therapy work in treating patients with stage IIIC-IV serous uterine cancer. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, stopping them from dividing, or stopping them from spreading. Giving the drugs in different ways may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy followed by radiation therapy may be an effective treatment for uterine cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity (as defined by National Cancer Institute [NCI] Common Toxicity Criteria version [v.] 4.0) of weekly intravenous (IV) paclitaxel with intraperitoneal (IP) carboplatin chemotherapy given every third week, followed by radiation therapy (RT) in patients with advanced stage uterine serous cancer (USC).

II. To determine the feasibility of this regimen in women with advanced stage USC.

SECONDARY OBJECTIVES:

I. To assess the frequency and the reasons for early discontinuation of the study treatments.

II. To describe patient-reported quality of life parameters at specified time points during the study using validated questionnaires: European Organization for Research and the Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 and QLQ-ovarian cancer module (OV)28.

TERTIARY OBJECTIVES:

I. To define patterns of recurrence (e.g. local versus distant) and progression-free survival in patients with advanced and recurrent USC treated with dose dense IV paclitaxel and IP carboplatin therapy.

II. To correlate surrogate endpoint biomarkers that is performed in standard histology processing (estrogen receptor and progesterone receptor status as well as human epidermal growth factor 2 [Her2/neu] status) with progression-free survival and prognosis.

III. To assess the potential late effects of combined intraperitoneal chemotherapy and radiotherapy on the gastrointestinal, genitoureteral, bone marrow and other body systems beginning at 6 months post treatment completion during routine office visits.

OUTLINE:

CHEMOTHERAPY: Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15 and carboplatin intraperitoneally (IP) on day 1. Treatment repeats every 21 days for up to 6 courses (weeks 1-18) in the absence of disease progression or unacceptable toxicity.

RADIATION: At provider discretion, patients may undergo 3-dimensional (3D) conformal or intensity-modulated radiation therapy (IMRT) 5 days a week for 5 weeks (weeks 19-23).

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then yearly thereafter for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytologically documented primary International Federation of Gynecology and Obstetrics (FIGO) stage 3C1, 3C2, stage 4A, and 4B uterine serous carcinoma; in addition, certain stage 3A and B disease are also allowed

  * Residual disease after primary surgery:

    * Eligible:

      * Stage 3A and B (pelvic, but confined to adnexa or vagina), residual disease present
      * Stage 3CI (pelvic node positive)
      * Stage 3CII (para-aortic node positive)
      * Stage 4A (bladder or pelvic bowel)
      * Stage 4B (distant metastases [mets] including abdominal mets), completely resected
    * Not eligible

      * Stage 3A and B (pelvic, but confined to adnexa or vagina), completely resected
      * Stage 4B (distant mets including abdominal mets), residual disease present
* All patients must have a procedure for determining diagnosis of high-risk uterine cancer (HRUC); minimum surgical intervention required is tissue biopsy (may be from endometrium), if significant clinical evidence exists to support a stage 3 or 4 diagnosis; as per the discretion of the surgeon, complete surgical staging should include: total abdominal hysterectomy, bilateral salpingo-oophorectomy, peritoneal washings, omental biopsy and lymph node samplings; this is typically the standard unless the disease is bulky or the clinician feels the patient would be best served by chemotherapy and radiation therapy after histologic diagnosis is confirmed
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Written voluntary informed consent

Exclusion Criteria:

* Distant metastasis to the lung, bone or brain; typically, most stage 4 uterine papillary serous cancer (UPSC) is confined to the abdomen on presentation
* Serum glutamic oxaloacetic transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) > 2.5 times the institutional upper limit of normal (ULN)
* Total serum bilirubin > 1.5 mg/dl
* Serum creatinine > 2.0 mg/dl
* Platelets < 100,000/mm^3
* Absolute neutrophil count (ANC) < 1500/mm^3
* Hemoglobin < 8.0 g/dl (the patient may be transfused prior to study entry)
* History of abdominal/pelvic radiation therapy
* Severe or uncontrolled, concurrent medical disease (e.g. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.)
* Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at the time of study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Frimer, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled into the study between. The 1st participant was enrolled on 4/10/2014 and the final participant was enrolled into the study on 4/5/2016. No further participants have been enrolled since April 2016.
Pre-assignment Details: 4 participants consented but only 3 were enrolled. One participant failed screening due to the onset of an adverse event.
Groups:
- Treatment (Paclitaxel, Carboplatin, Radiotherapy): CHEMOTHERAPY: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IP on day 1. Treatment repeats every 21 days for up to 6 courses (weeks 1-18) in the absence of disease progression or unacceptable toxicity.
  RADIATION: At provider discretion, patients may undergo 3D conformal or IMRT 5 days a week for 5 weeks (weeks 19-23).
  Paclitaxel: Given IV
  Carboplatin: Given Intraperitoneal (IP)
  3-Dimensional Conformal Radiation Therapy: Undergo 3D conformal radiation therapy
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  Quality-of-Life Assessment: Ancillary studies
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
Started | 3
Completed | 1
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 4 participants were consented but only 3 participants were enrolled into the study. One participants screen failed shortly after consent due to the onset of and adverse event. Baseline demographics provided for all 4 participants.
Groups:
- Treatment (Paclitaxel, Carboplatin, Radiotherapy): CHEMOTHERAPY: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IP on day 1. Treatment repeats every 21 days for up to 6 courses (weeks 1-18) in the absence of disease progression or unacceptable toxicity.
  RADIATION: At provider discretion, patients may undergo 3D conformal or IMRT 5 days a week for 5 weeks (weeks 19-23).
  Paclitaxel: Given IV
  Carboplatin: Given IP
  3-Dimensional Conformal Radiation Therapy: Undergo 3D conformal radiation therapy
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  Quality-of-Life Assessment: Ancillary studies
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Degree of Tolerability, Estimated by the Proportion of Participants Who Complete 6 Treatment Cycles of IP Carboplatin
Description: At the end of the study, the proportion of patients who tolerated the therapy will be estimated, along with corresponding 95% confidence intervals. Reasons for discontinuation of therapy will be categorized and summarized by computing frequencies.
Time Frame: Up to 18 weeks
Population: Data was not collected/aggregated and therefore not analyzed for Degree of Tolerability
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival
Description: The proportion of responders at one year will be estimated with the Kaplan-Meier method. Surrogate endpoint biomarkers including estrogen, progesterone, and Her2/neu receptor status will be correlated with progression-free survival using the Cox Proportional Hazards model, provided the availability of a sufficient number of events.
Time Frame: The duration of time from start of treatment to time of progression, or death, whichever happens first, assessed at 1 year
Population: Data was not collected/aggregated and therefore not analyzed for Progression Free Survival
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Minimally upon completion of radiation therapy at 26 weeks after treatment initiation. Further adverse event evaluations as clinically indicated.
Description: 4 participants were consented but only 3 participants were enrolled into the study. One participants screen failed shortly after consent due to the onset of and adverse event. Baseline demographics provided for all 4 participants.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Radiotherapy) (N=4)
Hematuria (Renal and urinary disorders) | 1 (1)
Neutropenia (febrile) (Blood and lymphatic system disorders) | 1 (2) — Grade 4. Study drug interrupted both times
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Radiotherapy) (N=4)
Fatigue (General disorders) | 1 (1) — Grade 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) — Grade 1
Weight Loss (Investigations) | 1 (2) — Grades 1-2
Constipation (Gastrointestinal disorders) | 1 (1) — Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1
Anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Grade 1
Peripheral Neuropathy (Nervous system disorders) | 1 (1) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No